CLINICAL TRIAL: NCT02863393
Title: Intentional Diaphragmatic Breathing Exercise Improves the Metabolic Profiles of Patients With Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Diaphragmatic Breathing Exercise Improves Non-alcoholic Fatty Liver Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Couldnt find sponor for this study
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N201603004
Record Dates: First submitted 2016-06-28; First posted 2016-08-11 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-04

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diaphragmatic breathing exercise (Experimental): The aim of this study is to ameliorate hepatic inflammation by using diaphragmatic breathing exercises instead of aerobic exercise to reduce the fat in liver inflammation.
  Interventions: Other: Diaphragmatic breathing exercise

INTERVENTIONS:
Other: Diaphragmatic breathing exercise — Through diaphragmatic breathing exercise to verify the impact of this item interventions on patients' metabolism indicators.

SUMMARY:
The non-alcoholic fatty liver disease is increasing and associated with obesity, diabetes and hyperlipidemia in recent years. Aerobic exercise indeed reduces adipose, hepatic insulin resistance and hepatic fat. However, diaphragmatic breathing improves cardiopulmonary function, the oxygen content of the body and therefore reduces inflammation of cells. The aim of this study is to ameliorate hepatic inflammation by using diaphragmatic breathing exercises instead of aerobic exercise to reduce the fat in liver inflammation.

DETAILED DESCRIPTION:
The non-alcoholic fatty liver disease is increasing and associated with obesity, diabetes and hyperlipidemia in recent years. Aerobic exercise indeed reduces adipose, hepatic insulin resistance and hepatic fat. However, diaphragmatic breathing improves cardiopulmonary function, the oxygen content of the body and therefore reduces inflammation of cells. The aim of this study is to ameliorate hepatic inflammation by using diaphragmatic breathing exercises instead of aerobic exercise to reduce the fat in liver inflammation. The project intends to be accomplished within three years because of the ideal exercise leaves an uncertain question for curing non-alcoholic fatty liver disease. Hence, with the literature and empirical data analysis to review and identify the strength of patients' motion and duration, carry out a pilot observational study by including 20 patients, then teach diaphragmatic breathing exercises in the first year of the project. Observe the initial correlation measurement, the variables of the following one month and three months. For the second year, develop the training of diaphragmatic breathing process with assisting device (Diaphragmatic breathing-facilitated exercise device). Use diaphragmatic breathing exercise assisting device in a 12-week program of diaphragmatic breathing on randomized clinical trial, verifying the impact of this item interventions on patients' metabolism indicators in the final year.The project includes people who are over 20 years old without the non-alcoholic fatty liver disease. Taking liver function, body mass index, the thickness of subcutaneous fat, heart rate variability, metabolism indicators are mainly study measured variables. Regression Analysis helps understand the correlation between breathing exercise and indicators related to the disease. With the intervention of diaphragmatic breathing assist device, the program extensions to the two-factor analysis of variance (two-way ANOVA) as the results of verification. The study results can provide a reference for clinicians, thereby improving the prognosis of non-alcoholic fatty liver disease people.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are confirmed by echo without non-alcoholic fatty liver disease and over 20 year-old, and willing to learn the exercise.

Exclusion Criteria:

* Patients who could drop out the trial if he or she doesn't want to continue the exercise.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
AST and ALT | Up to 3 months to collect data

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shun Wu, Doctor, Study Director — Wanfang Hospital

IPD SHARING:
Plan to Share IPD: No